CLINICAL TRIAL: NCT02973932
Title: Internet-based Cognitive Behavioral Psychotherapy for Children and Adolescents With Obsessive-compulsive Disorder
Brief Title: iCBT for Children and Adolescents With Obsessive-compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, PD Dr. Annette Conzelmann, PD Dr. Annette Conzelmann, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F.1331477
Record Dates: First submitted 2016-11-07; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Psychotherapy Intervention Evaluation
Keywords: cognitive-behavioral psychotherapy; obsessive-compulsive disorder; internet-based
MeSH Terms: conditions — Obsessive-Compulsive Disorder

ARMS (1):
- Internet-based psychotherapy (Experimental)
  Interventions: Behavioral: Cognitive-bahavioral psychotherapy

INTERVENTIONS:
Behavioral: Cognitive-bahavioral psychotherapy

SUMMARY:
Internet-based psychotherapy for children and adolescents with obsessive-compulsive symptoms and an age of 7 to 17 years. Sessions are verified with teleconferencing with an psychotherapist, children and their parents. The psychotherapy is supported by an App and a wristband to obtain psychophysiological data.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (ages 7-17) with a primary DSM-5 obsessive-compulsive disorder and at least 1 primary caretaker
* German-speaking (child & caretakers)
* Family home equipped with broadband connection and appropriate computer, monitor, HD webcam, and speaker and smart phone

Exclusion Criteria:

* IQ below 70
* A psychiatric comorbidity that makes participation clinically inappropriate (for example, primary anorexia nervosa), depression with suicidality that requires acute treatment, and psychosis

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The Schedule for Affective Disorders and Schizophrenia for School-Age Children Present and Lifetime Version (K-SADS-PL) | beginning of the study and end therapy (about 16 weeks)
The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | beginning of the study and end therapy (about 16 weeks)
Children's Global Assessment Scale (CGAS) | beginning of the study and end therapy (about 16 weeks)
Child Behavior Checklist (CBCL) | beginning of the study and end therapy (about 16 weeks)
Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents (KINDL) | beginning of the study and end therapy (about 16 weeks)
Impairment by OCD symptoms | Every day throughout the therapy process (14 weeks)
  assessed by App
Extend of avoidance behavior | Every day throughout the therapy process (14 weeks)
  assessed by App
Daily mood | Every day throughout the therapy process (14 weeks)
  assessed by App
How the day was | Every day throughout the therapy process (14 weeks)
  assessed by App
How strong OCD is | Every week throughout the therapy process (14 weeks)
  assessed by App
How Every week throughout the therapy processgood e progress was with specific treatment goals | Every week throughout the therapy process (14 weeks)
  assessed by App
Anxiety ratings during exposures | Every week three days beginning with session 4 up to 14
  assessed by App
Heart rate variability | Every day throughout the therapy (14 weeks)
  assessed with wristband
Skin conductance level | Every day throughout the therapy (14 weeks)
  assessed with wristband
Body temperature | Every day throughout the therapy (14 weeks)
  assessed with wristband
Body movements | Every day throughout the therapy (14 weeks)
  assessed with wristband

CONTACTS AND LOCATIONS:
Overall Officials: Annette Conzelmann, PhD, Principal Investigator — Department of Child and Adolescent Psychiatry University of Tübingen